CLINICAL TRIAL: NCT01559077
Title: A Phase 1, Randomized, Single-blind, Placebo-Controlled, Single Ascending Dose, Safety, Tolerability and Pharmacokinetics Study of ALN-TTR02 in Healthy Volunteers
Brief Title: Trial to Evaluate Safety, Tolerability, and Parmacokinetics of ALN-TTR02 in Healthy Volunteer Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-TTR02-001
Record Dates: First submitted 2012-03-19; First posted 2012-03-21 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: TTR-mediated Amyloidosis
Keywords: ATTR
MeSH Terms: interventions — patisiran

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-TTR02 (Active Comparator)
  Interventions: Drug: ALN-TTR02
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-TTR02 — Dose levels between 0.01 and 0.5 mg/kg by intravenous (IV) infusion
  Arms: ALN-TTR02
Drug: Sterile Normal Saline (0.9% NaCl) — Calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of a single dose of ALN-TTR02 in healthy volunteer subjects.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index must be between 18.0 kg/m2 and ≤ 31.5 kg/m2;
* Non-smokers for at least 3 months preceding screening;
* Females subjects must be of non-childbearing potential e.g., post-menopausal or pre-menopausal with surgical sterilization;
* Males agree to use appropriate contraception;
* Medical history must be verified by either a personal physician or medical practitioner as appropriate;
* Willing to give written informed consent and are willing to comply with the study requirements.

Exclusion Criteria:

* Known hepatitis B surface antigen (HBsAg), hepatitis B virus (HBV), hepatitis C virus (HCV) or human immunodeficiency virus (HIV) infection
* Multiple drug allergies or know sensitivity to oligonucleotide
* History of drug abuse and/or alcohol abuse
* Receiving an investigational agent within 3 months prior to study drug administration
* Subjects with safety laboratory test results deemed clinical significant by the Investigator;
* Received prescription drugs within 4 weeks of first dosing
* Subjects who have donated more than 500 mL of blood within the 3 months prior to ALN-PCS02 or placebo administration;
* Subjects who have used prescription drugs within 4 weeks of first dosing
* Considered unfit for the study by the Principal Investigator
* Employee or family member of the sponsor or the clinical study site personnel

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2012-03; Primary Completion 2012-06 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs) and study drug discontinuation. | Up to 28 days

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of ALN-TTR02 (Cmax, tmax, t1/2, AUC0-last, CL). | Up to 180 days
Effect of ALN-TTR02 on transthyretin (TTR), vitamin A, and retinol binding protein (RBP) (Determination of % Lowering of TTR, vitamin A and RBP to pretreatment/Baseline Levels) | Up to 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Jared Gollob, MD, Study Director — Alnylam Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Clinical Site, Leeds
  - Clinical Site, London

REFERENCES:
- [Derived] Coelho T, Adams D, Silva A, Lozeron P, Hawkins PN, Mant T, Perez J, Chiesa J, Warrington S, Tranter E, Munisamy M, Falzone R, Harrop J, Cehelsky J, Bettencourt BR, Geissler M, Butler JS, Sehgal A, Meyers RE, Chen Q, Borland T, Hutabarat RM, Clausen VA, Alvarez R, Fitzgerald K, Gamba-Vitalo C, Nochur SV, Vaishnaw AK, Sah DW, Gollob JA, Suhr OB. Safety and efficacy of RNAi therapy for transthyretin amyloidosis. N Engl J Med. 2013 Aug 29;369(9):819-29. doi: 10.1056/NEJMoa1208760. PMID 23984729